CLINICAL TRIAL: NCT05371418
Title: Controlled Split Mouth Study of Effect of Orthodontic and Guided Bone Regeneration on Angular Bone Loss of Over-erupted Tooth
Brief Title: Comparative Clinical and Radiographical Evaluation of Treatment of Angular Bone Defect Related to Over Erupted Tooth Using GTR Followed by Orthodontic Intrusion Versus Orthodontic Intrusion Followed by GTR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, rehab ghouraba, principle investigator, Tanta University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3333
Record Dates: First submitted 2022-01-12; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Bone Loss; Occlusion
Keywords: overerupted tooth; angular bone loss; orthodontic intrusion
MeSH Terms: conditions — Bone Diseases, Metabolic; Bites and Stings | interventions — Surgical Procedures, Operative; Guided Tissue Regeneration

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- guided regeneration (GTR) followed by orthodontic intrusion (Experimental): Ten over erupted teeth were selected with an angular bone loss with presence of their opposing for spilt mouth study aged from 20- 35 years old, were treated by GTR followed by Orthodontic intrusion
  Interventions: Procedure: surgical (guided tissue regeneration)
- Orthodontic intrusion followed by GTR (Experimental): Ten over erupted teeth were selected with an angular bone loss with presence of their opposing for spilt mouth study aged from 20- 35 years old, were treated by orthodontic intrusion followed by GTR
  Interventions: Device: orthodontic intrusion followed by guided tissue regeneration GTR

INTERVENTIONS:
Procedure: surgical (guided tissue regeneration) — In group 1 (G1), ten teeth over erupted with angular bone loss were treated by guided tissue regeneration (GTR) followed by Orthodontic intrusion
  Other Names: guided tissue regeneration
  Arms: guided regeneration (GTR) followed by orthodontic intrusion
Device: orthodontic intrusion followed by guided tissue regeneration GTR — . In group 2 (G2), ten teeth over erupted with angular bone loss were treated by Orthodontic intrusion (OI) followed by guided tissue regeneration (GTR)
  Other Names: orthodontic intrusion
  Arms: Orthodontic intrusion followed by GTR

SUMMARY:
Occlusal prematurity leading to loss of vertical stopping points between teeth can lead to teeth over eruption creating abnormal contact area which favors food accumulation and plaque retention. All these factors can lead to gingival inflammation and bone loss which may be worsen by abnormal occlusal force. Thus, orthodontic evaluation and treatment with periodontic therapy is mandatory to achieve proper treatment.

Aim of the work: To evaluate and compare clinically and radiographically between effect of guided tissue regeneration (GTR) followed by orthodontic intrusion versus orthodontic intrusion followed by GTR in treatment of over erupted tooth with angular bone loss

DETAILED DESCRIPTION:
Abstract Occlusal prematurity leading to loss of vertical stopping points between teeth can lead to teeth over eruption creating abnormal contact area which favors food accumulation and plaque retention. All these factors can lead to gingival inflammation and bone loss which may be worsen by abnormal occlusal force. Thus, orthodontic evaluation and treatment with periodontic therapy is mandatory to achieve proper treatment.

Aim of the work: To evaluate and compare clinically and radiographically between effect of guided tissue regeneration (GTR) followed by orthodontic intrusion versus orthodontic intrusion followed by GTR in treatment of over erupted tooth with angular bone loss Material and methods: Twenty teeth in ten cases were selected with at least two teeth with vertical over eruption and angular bone loss with presence of their opposing for spilt mouth study aged from 20- 35 years old. In group 1 (G1), ten teeth over erupted with angular bone loss were treated by GTR followed by Orthodontic intrusion whereas, in group two (G2) ten teeth over erupted with angular bone loss were treated by orthodontic intrusion followed by GTR. All cases were evaluated clinically for pocket depth (PD), bleeding on probing (BOP), tooth mobility prior starting phase one therapy, at re-evaluation and at six- and 12-months post starting either GTR or orthodontic intrusion. Also, radiographical evaluation was assessed using CBCT scan at end of re-evaluation, at six- and 12-months post starting either GTR or orthodontic intrusion to evaluate amount of orthodontic intrusion, amount of change of bone area and length related to angular defect in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Over erupted tooth with angular bone loss with presence of opposing
* Mobility doesn't exceed grade two
* No gingival recession more than 3mm

Exclusion Criteria:

* Systematic diseases that complicate oral surgery such as hyperparathyroidism, bleeding disorders,....etc.
* Smokers
* Patients with negative attitude towards oral hygiene

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-10-11 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
the effect of GTR followed by OI in G1and OI followed by GTR in G2 evaluated clinically regarding pocket depth and tooth mobility | 12-15 months
  pocket depth will be measured by mm, and tooth mobility with giving scoreM0: Physiological mobility,M1: Slightly increased mobility,M2: Definitive considerable increase in mobility but no impairment of function, M3: Extreme mobility, loose tooth that would be incompatible in function.
  these measurements were done prior starting phase one, one month after finishing phase one (Re-evaluation phase) and at six- and 12-months post starting either GTR or orthodontic intrusion (OI)
the effect of GTR followed by OI in G1and OI followed by GTR in G2 evaluated radiographically by cone beam computed tomography (CBCT) regarding bone defect area bymm2 and defect area dimensional changes by mm2 | 12-15 months
  the defect area was measured by mm2 at re-evaluation phase, 6 months post GTR in G1 or OI in G2 and after one year from re-evaluation phase in both groups and defect area dimensional changes by mm2 which was evaluated by subtracting value of bone area at 6 months post GTR in G1 or OI in G2 from bone area at Re-evaluation and and subtracting bone area at one year from re-evaluation from bone area at 6 months post GTR in G1 or OI in G2

SECONDARY OUTCOMES:
the effect of GTR followed by OI in G1and OI followed by GTR in G2 evaluated clinically regarding bleeding upon probing | 12-15 months
  All cases were evaluated clinically for bleeding upon probing (BOP) for score (0) healthy gingiva; no bleeding upon insertion of periodontal probe interproximal, (1) edematous, reddened gingiva; no bleeding upon insertion of periodontal probe interproximal, (2) bleeding without flow upon periodontal probe interproximal, (3)bleeding with flow along gingival margin upon insertion of periodontal probe interproximal (4)copious bleeding upon insertion of periodontal probe interproximal and (5) severe inflammation, marked redness and . These measurements were done prior starting phase one, one month after finishing phase one (Re-evaluation phase) and at six- and 12-months post starting either GTR or orthodontic intrusion (OI)
the effect of GTR followed by OI in G1and OI followed by GTR in G2 evaluated radiographically using CBCT regarding defect depth | 12-15 months
  the defect depth was measured by mm at re-evaluation phase, 6 months post GTR in G1 or OI in G2 and after one year from re-evaluation phase in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Rehab F Ghouraba, PHD, Principal Investigator — Tanta University
Locations (1):
- Rehab Fouad Ghouraba, Tanta, Grabia, Egypt